CLINICAL TRIAL: NCT01935232
Title: Validation of Bindex Bone Ultrasonometer for Osteoporosis Diagnostics
Brief Title: Bindex Ultrasonometer for Osteoporosis Diagnostics
Status: Terminated | Type: Observational
Why Stopped: Institution not able to carry out research as of 2015
Sponsor: Bone Index Finland Ltd (Industry)
Collaborators: HealthEast Care System (Other)
Responsible Party: Sponsor
Other Study IDs: Bind01; BoneIndex01 (Other: Bone Index Finland Ltd.)
Record Dates: First submitted 2013-08-21; First posted 2013-09-05 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Osteoporosis
Keywords: Osteoporosis, diagnostics, ultrasound
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Men: 140 Men
- Female: 500 Female

SUMMARY:
Osteoporosis is a disease that leads to impaired skeletal strength and increased fracture risk. Among 200 million osteoporotic patients (Tarantino, Cannata et al. 2007) most are diagnosed only after a fracture. We expect with our aging population to see a significant increase in the prevalence of osteoporosis. It is estimated that over 75% of osteoporotic patients are not diagnosed and do not receive treatment for their condition.

This research plan describes a study for clinical validation of the novel ultrasound device (Bindex®, Bone Index Finland Ltd.). In a preliminary study, the technique has been validated in a Finnish postmenopausal woman population of 285 healthy and 56 osteoporotic subjects (n = 341 in total). Significant and good correlation was observed between Density Index (DI) determined with Bindex and femoral neck bone mineral density determined with DXA (r = 0.65 - 0.70). In addition, with determination of 90% sensitivity and specificity thresholds, significant number (65-75%) of patients could be diagnosed without additional verification with DXA.

For validation of the technique in US population, our study plan is presented for determination of diagnostic thresholds for osteoporosis. Taken together, DI with Bindex, lumbar spine and femoral bone BMD with DXA are obtained from 500 postmenopausal women and 140 men. The study will be carried out at the HealthEast Osteoporosis Care service in Woodbury, MN.

1. To investigate the capability of DI for prediction of proximal femur and lumbar spine BMD;
2. To develop national diagnostic thresholds for DI in prediction of osteoporosis status with a reference population (American-Caucasian) of 500 (if prevalence of osteoporosis is 20%) post-menopausal females (50-90 years);
3. To investigate ability of Density Index + FRAX with BMI in fracture risk prediction;
4. To investigate correlation between lumbar spine or proximal femur BMD and Density Index in 140 men at wide age range (20-90 years), 70 with osteoporosis and 70 with normal or low bone mass. Determine diagnostic thresholds for DI in men.

DETAILED DESCRIPTION:
Quality

On-site training for the ultrasound device will be provided. Reproducibility shall be determined for each operator. After 100 patient have been measured, data shall be analysed, validated for value ranges and for consistency with other data fields in registry. Assessment of possible missing data fields. If measurement related, corrective and preventive actions shall be taken prior continuation of the study.

Data Registry

Data will be collected at the time of the bone density and ultrasound (DI) exams. Information collected will be entered into a database for statistical analysis. In addition to patient characteristics, 7 questions shall be presented to each patient to gather fracture risk related data (http://www.shef.ac.uk/FRAX):

1. Previous fracture
2. Parent fip fracture
3. Current smoking
4. Use of Glucocorticoids
5. Rheumatoid arthritis
6. Secondary osteoporosis
7. Alcohol 3 or more units/day

Confidentiality

1. Any of the data from this study will not be a part of permanent record (identifiable to the subject) that will be made available to physician, employer, supervisor, student, FDA, etc.
2. Data will be kept in paper form indefinitely at HealthEast Osteoporosis Care. All research data is kept in locked cabinetry.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women and men referred for bone density examination.

Exclusion Criteria:

* Patients unable to sign consent for participation.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: American-Caucasian female (n=500) American-Caucasian men (n=140)
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Threshold values for DI to reach 90% sensitivity and specificity with the method in diagnostics of Osteoporosis. | 1 year

SECONDARY OUTCOMES:
Amount subjects that can be diagnosed with the established thresholds for DI. Amount of subjects that would require additional examination to verify diagnosis.Correlation between BMD at neck, total hip and lumbar spine with DI. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Christine Simonelli, MD, Principal Investigator — HealthEast Osteoporosis Care; Janne P Karjalainen, PhD, Study Director — Bone Index Finland Ltd; Ossi Riekkinen, PhD, Study Director — Bone Index Finland Ltd
Locations (1):
- HealthEast Clinic, Saint Paul, Minnesota, United States